CLINICAL TRIAL: NCT03772496
Title: A Multicenter, Double-blind, Prospective Cohort Study of Diagnostic Significance of Circulating Tumor Cells in Patients With Thyroid Nodules
Brief Title: Diagnostic Significance of CTCs in Patients With Thyroid Nodules (Circulating Tumor Cells)
Acronym: CTCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, liu jie, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S0006YIO
Record Dates: First submitted 2018-11-23; First posted 2018-12-11 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Nodule; Diagnoses Disease
Keywords: fine needle aspiration biopsy; Circulating tumor cells; benign; malignant
MeSH Terms: conditions — Thyroid Nodule; Neoplastic Cells, Circulating | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- circulating tumor cells (Experimental): circulating tumor cells test and FNAB will be performed at the same time
  Interventions: Diagnostic Test: circulating tumor cells test; Diagnostic Test: Fine needle aspiration biopsy

INTERVENTIONS:
Diagnostic Test: circulating tumor cells test — 10 ml Peripheral blood are drawn from patients enrolled before surgery/FNAB and centrifuged to collect the peripheral blood mononuclear cells. Then, negative and positive immunomagnetic selections are used to exclude white blood cells and enrich tumor cells. After isolating mRNA, RT-PCR array is used to measure expression of target genes.
Diagnostic Test: Fine needle aspiration biopsy — patients with potential malignant thyroid nodules are performed fine needle aspiration biopsy with the aid of ultrasound. The result of FNAB were classified by Bethesda rating system.

SUMMARY:
Thyroid nodule patients with suggestion of fine needle aspiration biopsy (FNAB) offered by ultrasound are enrolled in the study. CTCs tested by Optimizing method and FNAB will be performed simultaneously. This is a double blind trial which pathologists and inspectors of CTCs don't know the result of each other. Surgical pathology and diagnostic results of FNAB is the primary endpoint and comparison will be made to see if CTCs combined with ultrasound can get similar diagnostic performance as FNAB. The diagnostic results of FNAB included Bethesda class II and more than V which are defined as benign and malignant, respectively.

DETAILED DESCRIPTION:
Some retrospective analysises showed CTCs is considered to be valuable for diagnosis, staging, prognosis and follow-up in several types of cancers and some mRNA markers are helpful in differentiating patients with benign versus malignant thyroid disease. However, the lack of sensitivity and specificity of mRNA measurements restricted their clinical application. The aim of this study is to see if optimizing test method combined with ultrasound can get similar diagnostic performance. 200 patients with thyroid nodules (≤2cm) which need to undergo FNAB will be enrolled in four centers of northern China. Patients will simultaneously undergo CTCs tests and FNAB. And following treatments will be performed according to the previous standard. Allowed by the patients, the investigators will obtain 10ml peripheral blood samples from the participants to make a CTCs test before any FNAB. The primary end point is the pathologically confirmed benign versus malignant thyroid disease, which including surgical pathology and diagnostic results of FNAB.

ELIGIBILITY:
Inclusion Criteria:

* patients with thyroid nodules (≤2cm) untreatment FNAB suggested by ultrasound

Exclusion Criteria:

* the history of other cancer the history of thyroid surgery Bethesda class 3 without surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
post-operative pathology | 10 days after surgery
  Patients with malignant results of FNAB (Bethesda V and VI)non-diagnostic results of FNAB (Bethesda class I , III, IV)will be suggested to undergo surgery. Those patients who underwent surgery are enrolled in our study and are performed a post-operative pathology, which have a higher evidence rank than FNAB. According to post-operative pathology, any type of thyroid carcinoma is defined as malignant, and patients who have not been strong enough to be diagnosed with carcinoma is defined as benign disease.
diagnostic results of FNAB | 10 days after FNAB
  The result of FNAB are classified by Bethesda rating system. Bethesda class I is considered the sample is not qualified, Bethesda class II is defined as benign, Bethesda class III and IV are defined as non-diagnostic result, which need further verified by surgery.Bethesda class V and VI are defined as malignant.

CONTACTS AND LOCATIONS:
Overall Officials: jie liu, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No